CLINICAL TRIAL: NCT03122444
Title: A Pre-Surgical Window of Opportunity Trial Investigating the Effect of Imipramine on Previously Untreated Breast Cancer (CTMS# 17-0037)
Brief Title: Imipramine on ER+ve and Triple Negative Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Virginia G. Kaklamani, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 17-0037
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Imipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imipramine (Experimental): Imipramine will initially be 50mg and this will be increased by 50mg every other day as tolerated to 200 mg.
  Interventions: Drug: Imipramine

INTERVENTIONS:
Drug: Imipramine — Imipramine will be given daily for 21-30 days.

SUMMARY:
Comparing changes in biomarkers from a diagnostic core needle biopsy to surgical pathology specimen or repeat core needle biopsy.

DETAILED DESCRIPTION:
This will be a single arm, non-randomized, pre-surgical clinical trial of women with newly diagnosed triple negative breast cancer comparing changes in biomarkers from a diagnostic core needle biopsy to surgical pathology specimen or repeat core needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Participants may be female or male who are 18 years old or older.
* Ability to consent to treatment - patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* Previously untreated breast cancer determined by a core needle biopsy showing invasive ductal carcinoma or invasive lobular carcinoma.
* A prior, unrelated, breast cancer is allowed.
* All breast cancers with possibility for surgical excision will be included.
* Patient must be able to take oral medications. Patients may not have any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study drug.
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test result within 14 days prior to the first dose of imipramine.
* Patients must be eligible for surgical resection of their breast cancer or repeat biopsy after completing treatment.
* Patients must have a complete history and physical examination within 30 days prior to registration.
* Patients must have a performance status of ECOG 0, 1, 2.
* Tissue block of initial biopsy specimen is available.
* Patient may not be concurrently enrolled in another investigational drug treatment study.

Exclusion Criteria:

* Known diagnosis of major depressive disorder, bipolar depression or psychosis
* ECOG 3 or 4
* Age >= 70 years
* Renal impairment defined as EGFR <30
* Hepatic impairment as judged by clinical investigator or bilirubin >2
* As judged by the investigator, severe uncontrolled concurrent medical conditions, psychiatric illness or social condition that would limit compliance with study requirements
* History of cardiac disease (arrhythmia, conduction abnormality, congenital prolonged QT syndrome, or prolonged QTc rhythm noted during initial EKG >480 ms)
* Current use of SSRI, SNRI, MAO inhibitor, tramadol or trazadone; or use of these agents within 14 days
* Inflammatory breast cancer
* Suicidal ideation or history of suicide attempt
* Myocardial infarction within 3 months of study initiation.
* Patients with Angle-Closure Glaucoma
* Pregnant or breast-feeding women. As there have been no well-controlled studies conducted with pregnant women to determine the effect of imipramine on the fetus. However, there have been clinical reports of congenital malformations associated with the use of the drug.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Decrease in the proliferation rate of triple negative breast cancer | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Virginia G Kaklamani, MD, Principal Investigator — Principal Investigator
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States